## The Safety and Efficacy of the Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) for Short Diagnostic Bronchoscopy Procedures

Statistical Analysis Plan
NCT03086408
June 9, 2020

Means and standard deviations were calculated for each of the patient characteristics. The statistical significance of differences between THRIVE and non-THRIVE patients was assessed using unpaired two sample Student's t-test with 95% confidence interval for all patient characteristics, without adjusting for multiple comparisons. For patients' gender, a chi-square test was used.